CLINICAL TRIAL: NCT05755815
Title: Ultrasound-guided Retrolaminar Block Versus Intraperitoneal Block for Postoperative Analgesia of Adult Patients Undergoing Laparoscopic Cholecystectomy: Randomized, Controlled Trial
Brief Title: Retrolaminar Block Versus Intraperitoneal Block for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amany Hazem abdelmaksood EL-deeb, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLB Block for cholecystectomy
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: retrolaminar block

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects and the resident assessing the outcomes will be blinded to the study group. A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation, perform the block, and administer bupivacaine solution.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (RLB block) (Active Comparator): Ultrasound-guided RLB block will be performed under strict aseptic precautions with patient turned to the lateral position.
  Interventions: Procedure: retrolaminar block
- Group B (Peritoneal block) (Active Comparator): Peritoneal block will be performed under strict aseptic precautions before giving an incision for the ports, and at the end of surgery and before the removal of trocars
  Interventions: Procedure: Peritoneal block

INTERVENTIONS:
Procedure: retrolaminar block — A high-frequency 12 MHz linear ultrasound probe will be used, patients will receive bilateral ultrasound-guided retrolaminar plane block with 20 mL of bupivacaine 0.25%. Their spines will be palpated from the vertebra prominens caudally to T7 and point will be marked to identify the spinous processes, which will be confirmed by ultrasound through counting from T12 with the characteristic last rib attached to its transverse process upward to the T7 lamina. The linear high frequency transducer (6-13 MHz) will be placed in the parasagittal plane one cm lateral to the midline. The needle will be inserted in the in-plane view of the ultrasound probe and will be advanced from downward to upward to target the T7 posterior lamina surface at an angle of 90˚ to the skin until the needle tip will be contacted the posterior surface of targeted lamina . After negative aspiration, 20 mL of bupivacaine 0.25% will be injected. The procedure was repeated following the same steps on the other side.
  Arms: Group A (RLB block)
Procedure: Peritoneal block — before giving an incision for the ports, 20 ml of 0.25% bupivacaine will be infiltrated subcutaneously over the port sites (6 ml will be infiltrated around each midline port site and 4 ml will be infiltrated around at the lateral port sites) and at the end of surgery and before the removal of trocars, 20 ml of 0.25% bupivacaine diluted in normal saline will be instilled by the surgeon intraperitoneally at gallbladder bed and under domes of both diaphragms under direct vision with a separate catheter passed through one of the trocars.. The pressure of the gas insufflation was kept within 10-12 mm Hg in all patients. At the end of surgery, CO2 was evacuated, and intraperitoneal anesthetic solution was left in situ.
  Arms: Group B (Peritoneal block)

SUMMARY:
Although laparoscopic cholecystectomy is a minimally invasive surgery, it causes moderate-severe pain. The aim of this study is to assess the quality of pain relief in patients who will undergo in laparoscopic cholecystectomy surgery receiving either retrolaminar block or peritoneal block by comparing and evaluating the differences between the two techniques. It is hypothesized that retrolaminar block will be comparable to peritoneal block as a promising effective alternative for analgesia for in laparoscopic cholecystectomy surgeries with fewer side effects.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) provides many advantages as less pain, shorter hospital stay, and earlier recovery, and it is a cost-effective procedure. Although it is a minimally invasive surgery, it causes moderate-severe pain. Pain has several sources but mostly visceral pain caused by tissue trauma during gall bladder resection is the most predominant component. Acute pain after laparoscopic cholecystectomy does not match pain after other laparoscopic surgeries because of its complexity, so proper management of pain should be procedure-specific and multimodal. Many analgesic interventions with different mechanisms have been studied for their effects on pain relief after laparoscopic cholecystectomy. Traditionally, opioids have been used to manage postoperative pain. However, an increasing awareness of opioid-related adverse events, including respiratory depression, paralytic ileus, and sedation, has led to a shift towards utilizing opioid-sparing techniques for postoperative analgesia. Ultrasound-guided retrolaminar block is a recent modified paravertebral technique for analgesia in thoracoabdominal procedures with a local anesthetic injected at the retrolaminar site. It has the advantage of being safe and easy compared with traditional thoracic epidural analgesia. It has a decreased incidence of complications such as hypotension, pleural disorder, and nerve injury.Intraperitoneal local anaesthetic administration has been used as a method for reducing postoperative pain. Intraperitoneal local anaesthetics acts on visceral nociceptors of peritoneum.Therefore, this study will be conducted to evaluate efficacy and safety of ultrasound guided retrolaminar block for postoperative analgesia in laparoscopic cholecystectomy surgery in comparison to intraperitoneal local anaesthetic administration.

Aim of the Study:

The aim of this study is to assess the quality of pain relief in patients who will undergo in laparoscopic cholecystectomy surgery receiving either retrolaminar block or peritoneal block by comparing and evaluating the differences between the two techniques. It is hypothesized that retrolaminar block will be comparable to peritoneal block as a promising effective alternative for analgesia for in laparoscopic cholecystectomy surgeries with fewer side effects.

Sample Size Calculation:

Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 11.0.4 for windows (2011) with time to first analgesic request as the primary outcome. Using the results published by ahmed et al 2021 with the mean time to first analgesic request in intraperitoneal instillation group was (2.88 ± 0.33 hours). Using a two-sided two-sample unequal-variance t-test., sample size of 54 patients is needed to achieve 90% power to detect 10 % difference in time to first analgesic request. Using a two-sided hypothesis test with a significance level of 0.05. A 10% drop out is considered, so a total of 60 patients will be enrolled (30 in each group) in this study

Methods:

The study will be conducted in Mansoura university hospital on sixty patients Who is Scheduled for laparoscopic cholecystectomy.They will be randomly assigned to two equal groups (retrolaminar group and peritoneal group) according to computer-generated table of random numbers using the permuted block randomization method. The group allocation will be concealed in sequentially numbered, sealed opaque envelopes which will be opened only after obtaining the written informed consent. Patient demographic data including age, sex and body weight will be recorded. A written informed consent will be obtained from all study subjects after ensuring confidentiality. The study protocol will be explained along with VAS to all patients after enrollment into the study. In both groups, the block will be under strict aseptic conditions after patient intubation and before skin incision.

Statistical Methods:

The collected data will be coded, processed, and analyzed using SPSS(Statistical Package for the Social Sciences) program (version 22) for Windows. Normality of numerical data distribution will be tested by Shapiro-Wilk test. Continuous data of normal distribution will be presented as mean ± SD (Standard deviation)and compared with the unpaired student's t test. Non-normally distributed data will be presented as median (range) and compared with the Mann-Whitney U test. Repeated measures ANOVA will be used for comparisons within the same group. Categorical data will be presented as number (percentage) and compared with the Chi-square test. All data will be considered statistically significant if P value is ≤ 0.05.Conditions

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) 1 or 2 patients.
* Scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Patient's refusal.
* Altered mental status or un-cooperative patients.
* History of known sensitivity to the used anesthetics.
* Bleeding or coagulation diathesis.
* Infection or redness at the injection site.
* Significant cardiac dysfunction, hepatic, or renal impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
First analgesic request | [Time Frame: Up to 24 hours after the procedure]
  The time of the first analgesic request for pethidine will be recorded.

SECONDARY OUTCOMES:
Visual analogue score (VAS) for pain assessment | Up to 24 hours after the procedure
  VAS score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) will be assessed every two hours for 24 hours after the procedure.
Total analgesic requirements of fentanyl | Up to 24 hours after the procedure
  The amount of pethidine consumption given as a rescue analgesia to patients will be measured all over the 24 hours.
Heart rate (HR) | Up to the end of the procedure
  HR will be recorded every 30min till the end of the procedure
Mean arterial pressure (MAP) | Up to the end of the procedure
  MAP will be recorded every 30min till the end of the procedure.
.Adverse effects | Up to 24 hours after the procedure
  Nausea, vomiting, hematoma, or allergic reactions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Amany H EL-Deeb, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bilge A, Basaran B, Et T, Korkusuz M, Yarimoglu R, Toprak H, Kumru N. Ultrasound-guided bilateral modified-thoracoabdominal nerve block through a perichondrial approach (M-TAPA) in patients undergoing laparoscopic cholecystectomy: a randomized double-blind controlled trial. BMC Anesthesiol. 2022 Oct 28;22(1):329. doi: 10.1186/s12871-022-01866-4. PMID 36307755
- [Result] Funk RD, Hilliard P, Ramachandran SK. Perioperative opioid usage: avoiding adverse effects. Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):32S-39S. doi: 10.1097/PRS.0000000000000680. PMID 25255004
- [Result] Gupta M, Naithani U, Singariya G, Gupta S. Comparison of 0.25% Ropivacaine for Intraperitoneal Instillation v/s Rectus Sheath Block for Postoperative Pain Relief Following Laparoscopic Cholecystectomy: A Prospective Study. J Clin Diagn Res. 2016 Aug;10(8):UC10-5. doi: 10.7860/JCDR/2016/18845.8309. Epub 2016 Aug 1. PMID 27656533
- [Result] Kamel AAF, Elhossieny KM, Hegab AS, Salem DAE. Ultrasound-guided Retrolaminar Block Versus Thoracic Epidural Analgesia for Pain Control Following Laparoscopic Cholecystectomy. Pain Physician. 2022 Sep;25(6):E795-E803. PMID 36122260
- [Result] Khandelwal H, Parag K, Singh A, Anand N, Govil N. Comparison of Subcostal Transversus Abdominis Block with Intraperitoneal Instillation of Levobupivacaine for Pain Relief after Laparoscopic Cholecystectomy: A Prospective Study. Anesth Essays Res. 2019 Jan-Mar;13(1):144-148. doi: 10.4103/aer.AER_3_19. PMID 31031495
- [Result] Mishra PK, Mani S, Singh RB. Evaluating the Efficacy of Pre-incisional Infiltration and Intraperitoneal Instillation of a Local Anesthetic Agent on Postoperative Analgesia and Hemodynamics in Patients Undergoing Laparoscopic Cholecystectomy Under General Anesthesia. Cureus. 2022 Mar 8;14(3):e22977. doi: 10.7759/cureus.22977. eCollection 2022 Mar. PMID 35415034
- [Result] Pizzi LT, Toner R, Foley K, Thomson E, Chow W, Kim M, Couto J, Royo M, Viscusi E. Relationship between potential opioid-related adverse effects and hospital length of stay in patients receiving opioids after orthopedic surgery. Pharmacotherapy. 2012 Jun;32(6):502-14. doi: 10.1002/j.1875-9114.2012.01101.x. Epub 2012 May 8. PMID 22570188